CLINICAL TRIAL: NCT03765437
Title: Safety of a Quadrivalent Influenza Vaccine (VaxigripTetra™) in Subjects Aged 6 Months and Older in Vietnam
Acronym: GQM10
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GQM10; U1111-1183-6274 (Other: UTN)
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: The study design is considered Phase 3 for the purpose of registration. This is a safety assessment study designed to provide safety data in Vietnamese participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quadrivalent Influenza Vaccine (Experimental): Quadrivalent Influenza Vaccine (split-virion, inactivated) Northern hemisphere seasonal formulation 2018-2019
  Interventions: Biological: Quadrivalent Influenza Vaccine

INTERVENTIONS:
Biological: Quadrivalent Influenza Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
  Other Names: VaxigripTetra™

SUMMARY:
The primary objective of this study is to describe the safety of the Quadrivalent Influenza Vaccine (QIV). Safety is assessed throughout the study period, and includes solicited injection site and systemic reactions (Day 0 to Day 7 post-vaccination); unsolicited adverse events up to Day 28, and serious adverse events occurring throughout the study.

DETAILED DESCRIPTION:
Study duration for previously unvaccinated participants aged 6 months to 8 years is approximately 56 days. Study duration for previously vaccinated participants aged 6 months to 8 years and any participant aged 9 years and older is approximately 28 days.

ELIGIBILITY:
Inclusion criteria :

* Aged 6 months and older on the day of inclusion
* Participants aged < 18 years: ICF has been signed and dated by the parent or another legally acceptable representative; Assent form has been signed and dated by the participant aged 12 to 15 years.
* Participants aged ≥ 16 years: ICF signed and dated by the participant.
* Participants are able to attend all scheduled visits and to comply with all study procedures. For participants aged 6 months to 17 years, parent/legally acceptable representative are able to attend all scheduled visits and to comply with all study procedures
* For participants < 2 years: Born at full term of pregnancy (≥ 37 weeks) and/or with a birth weight ≥ 2.5 kg

Exclusion criteria:

* Participant is pregnant, or lactating, or of childbearing potential and not using an effective method of contraception or abstinence from at least 4 weeks prior to vaccination until at least 4 weeks after vaccination. To be considered of non-childbearing potential, a woman must be pre-menarche or post-menopausal for at least 1 year, or surgically sterile
* Participation at the time of study enrollment (or in the 4 weeks preceding study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, device, or medical procedure
* Receipt of any vaccine in the 4 weeks preceding the study vaccination or planned receipt of any vaccine in the 4 weeks following the study vaccination.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Known systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substances
* Known thrombocytopenia, contraindicating intramuscular vaccination based on investigator's judgment
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating IM vaccination based on investigator's judgment
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness/body temperature (temperature ≥ 37.5 C or ≤ 35.5 C). A prospective subject should not be included in the study until the condition has resolved or the febrile event has subsided
* Identified as Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e. parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2019-03-17 (Actual); Study Completion 2019-03-17 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting solicited injection site reactions or systemic reactions | Within 7 days after vaccination
  Injection site reactions: tenderness/pain, erythema, swelling, induration, and haemorrhage.
  Systemic reactions: participants ≤ 23 months: fever, vomiting, crying abnormal, drowsiness, appetite lost, and irritability; participants 2 years and older: fever, headache, malaise, myalgia, and shivering.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Investigational Site Number 7040001, Việt Trì, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org